CLINICAL TRIAL: NCT00607867
Title: Metabolic Response to a LoBAG30 Diet in Diabetic Patients on Metformin
Brief Title: LoBAG30 Diet in Patients on Metformin
Acronym: LoBAG Diet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding ended before the study was completed.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-010-07F
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus; Diet
Keywords: Diabetes Mellitus (type 2); Diet; Glycohemoglobin; Lipids; Kidney Function; Glycemic Index; Dietary Protein; Dietary Carbohydrate
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): A LoBAG30, weight maintenance diet will be given to subjects on metformin. All food will be provided for 5 weeks.
  Interventions: Other: LoBAG30 diet
- Arm 2 (Placebo Comparator): A weight maintenance, control diet consisting of 55% carbohydrate, 15% protein, 30% fat will be given to subjects on metformin. All food will be provided for 5 weeks.
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: LoBAG30 diet — A LoBAG30 diet consists of 30% of total energy intake as carbohydrate, 30% protein, and 40% fat.
  Arms: Arm 1
Other: Control Diet — A control diet consists of 55% of total energy intake as carbohydrate, 15% protein, 30% fat
  Arms: Arm 2

SUMMARY:
We will determine the metabolic response to a Low Biologically Available Glucose Diet (LoBAG30) in subjects currently receiving the maximum dose of metformin as monotherapy in whom the glycohemoglobin is not at an acceptable level (>8.0%). Our hypothesis is that introduction of a LoBAG30 diet to subjects currently treated with a full therapeutic dose of metformin will improve blood glucose control in people who have not achieved an acceptable total glycohemoglobin on metformin alone.

DETAILED DESCRIPTION:
Subjects will ingest a control diet (55% carbohydrate (CHO), 15% protein, 30% fat) or a LoBAG30 diet (30% CHO, 30% protein, 40% fat) in a parallel design with block randomization in pairs of two. Subjects will return to the study center twice each week while on the diets to have blood glucose, glycohemoglobin, lactate, weight and blood pressure measured, and to have urine assayed for urea and creatinine. At the beginning and end of the 5 week study period, the subjects will be admitted to the study center for 28 hours during which time blood will be drawn for 24 hour profiles of glucose, insulin, other hormones and several metabolites. For those subjects randomized to the LoBAG30 arm of the study, the control diet will be given during the first 24 hour study period; the assigned diet will be given at the end of the 5 week period.

ELIGIBILITY:
Inclusion Criteria:

* People with type 2 diabetes mellitus who currently are receiving the maximal dose of metformin monotherapy (2500 mg/day).
* These subjects will have had a stable glycohemoglobin (tGHb) in an unacceptably high range (8-11%) for at least 4 months prior to beginning the study.
* Subjects with tGHB > 11% (HbA1c > 10%) will not be recruited into the study.

Exclusion Criteria:

* Hematological abnormalities
* liver disease
* kidney disease
* macroalbuminuria (>300 mg albumin/24 hours)
* untreated thyroid disease
* congestive heart failure
* angina
* life-threatening malignancies
* proliferative retinopathy
* severe diabetic neuropathy
* peripheral vascular disease
* serious psychological disorders
* a body mass index > 35
* and a fasting triglyceride of >400 mg/dl.

  * Subjects taking slow-release metformin will not be studied.
  * Subjects taking medications other than metformin, known to affect fuel metabolism such as:
* insulin
* the sulfonylureas
* glucagon-like peptide 1 (GLP-1) analogs and metabolic inhibitors
* pramlintide
* prednisone and similar steroids
* thyroid hormone
* antipsychotic medications
* thiazide diuretics
* medroxyprogesterone
* high dose aspirin, also will be excluded.

  * If concentrations of serum folate, B12 or iron are low, the subject will be excluded from the study until corrected, i.e. until normal concentrations are recorded.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gannon, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- VA Medical Center, Minneapolis, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Proposed study design was 20 subjects, 10/arm. (Parallel arm design requested by grant Reviewers.) At the end of the funding period, 14 subjects had been enrolled and studied, 7 in each arm.
Groups:
- LoBAG30 Diet: A LoBAG30, weight maintenance diet 30% CHO, 30% Pro, 50% fat
- Control Diet: A weight maintenance, control diet 55% CHO, 15% protein, 30% fat
Period: Overall Study
Arm/Group | LoBAG30 Diet | Control Diet
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with type 2 diabetes being treated with metformin
Groups:
- LoBAG30 Diet: A LoBAG30, weight maintenance diet 30% carbohydrate, 30% protein, and 40% fat.
- Control Diet: A weight maintenance, control diet consisting 55% carbohydrate, 15% protein, 30% fat
- Total: Total of all reporting groups
Arm/Group | LoBAG30 Diet | Control Diet | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Full Range); unit: years] | 62 [51 to 71] | 61 [53 to 66] | 61.6 [51 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in %Hemoglobin A1c at 5 Weeks From Baseline
Description: Hemoglobin A1c measured before and after 5 weeks on the diet
Time Frame: Baseline and 5 weeks after dietary intervention
Measure: Mean (Standard Error); unit: Change in % A1c at 5 weeks from baseli
Arm/Group | LoBAG30 Diet | Control Diet
Number analyzed (Participants) | 7 | 7
Change in % A1c at 5 weeks from baseli | -0.9 (0.23) | -0.9 (0.16)

2. Secondary Outcome: Microalbumin Excretion
Description: change in urinary albumin excretion was measured before dietary intervention and after 5 weeks of dietary intervention
Time Frame: baseline and 5 weeks after dietary intervention
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | LoBAG30 Diet | Control Diet
Number analyzed (Participants) | 7 | 7
mg/day | -0.9 (4.2) | -8.3 (3.5)

3. Primary Outcome: Change in Total Glucose Area at 5 Weeks From Baseline
Description: The area response is measured using zero as baseline. The area is measured before dietary intervention, and following 5 weeks of dietary intervention.
Time Frame: Baseline and 5 weeks after dietary intervention
Measure: Mean (Standard Error); unit: mg hr/dl
Arm/Group | LoBAG30 Diet | Control Diet
Number analyzed (Participants) | 7 | 7
mg hr/dl | -957 (302) | -691 (84)

4. Primary Outcome: Change in Body Weight at 5 Weeks From Baseline
Description: Subjects were to remain weight stable. We expected less than 2 pound weight change over 5 weeks. Weight was measured before dietary intervention, and after 5 weeks of dietary intervention.
Time Frame: baseline and 5 weeks after dietary intervention
Measure: Mean (Standard Error); unit: pounds
Arm/Group | LoBAG30 Diet | Control Diet
Number analyzed (Participants) | 7 | 7
pounds | -0.7 (0.7) | -2.6 (1.0)

5. Primary Outcome: Change in Overnight Fasting Glucose Concentration at 5 Weeks From Baseline
Description: Overnight fasting glucose concentration was measured before dietary intervention and after 5 weeks of dietary intervention.
Time Frame: baseline and 5 weeks after dietary intervention
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | LoBAG30 Diet | Control Diet
Number analyzed (Participants) | 7 | 7
mg/dl | -22 (16.5) | -33 (4.7)

6. Secondary Outcome: Change in Fasting Triglycerides at 5 Weeks From Baseline
Description: Overnight fasting triglycerides concentration was measured before dietary intervention and after 5 weeks of dietary intervention
Time Frame: baseline and 5 weeks after dietary intervention
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | LoBAG30 Diet | Control Diet
Number analyzed (Participants) | 7 | 7
mg/dl | -18 (12.9) | -24 (9.9)

ADVERSE EVENTS:
Groups:
- LoBAG30 Diet: A LoBAG30, weight maintenance diet will be given to subjects on metformin. All food will be provided for 5 weeks.
  LoBAG30 diet: A LoBAG30 diet consists of 30% of total energy intake as carbohydrate, 30% protein, and 40% fat.
- Control Diet: A weight maintenance, control diet consisting of 55% carbohydrate, 15% protein, 30% fat will be given to subjects on metformin. All food will be provided for 5 weeks.
  Control Diet: A control diet consists of 55% of total energy intake as carbohydrate, 15% protein, 30% fat
Arm/Group | LoBAG30 Diet | Control Diet
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Funding ended with only 14 subjects studied. With a parallel arm design, we were not able to draw any conclusions from the study. Funds were unavailable for a more sophisticated statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes